CLINICAL TRIAL: NCT01118143
Title: Effects of Communication Tailored to Oral Health Literacy Level of Adult Dental Patients: A Randomized Controlled Trial
Brief Title: Oral Health Literacy Tailored Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UIT/TkNN
Record Dates: First submitted 2010-04-28; First posted 2010-05-06 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-03

CONDITIONS: Periodontal Diseases; Dental Plaque; Dental Calculus; Sialorrhea; Streptococcal Infections; Lactobacillus Infection
MeSH Terms: conditions — Periodontal Diseases; Dental Plaque; Dental Calculus; Sialorrhea; Streptococcal Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention group (Experimental): Tailored oral health literacy instruction
  Interventions: Behavioral: Tailored oral health literacy instruction
- control group (No Intervention): Oral health instruction not tailored to oral health literacy level

INTERVENTIONS:
Behavioral: Tailored oral health literacy instruction — The intervention includes oral hygiene instruction tailored to the level of oral health literacy, and will include information about the outcome of the clinical examination. Providing relevant information to the participant will be in focus, and there will be given a personalized demonstration as well as guidance on how to conduct proper oral hygiene practices at home. The aim of the intervention is to improve oral hygiene and attitudes towards dental care by taking the literacy level of the participant into consideration.
  Other Names: Lifestyle counseling
  Arms: intervention group

SUMMARY:
The purpose of this study to investigate attitude, oral health literacy and psychological factors in order to evaluate if these factors are important for oral health in adults.

The hypotheses are:

* Multiple interactive demographic, and social and psychological factors contribute to the level of attitude and oral health literacy.
* There is an association between the level of oral health literacy and oral health status
* A structured intervention based on oral health literacy can change the attitude and improve the oral health status.
* Background knowledge has influence on attitude and oral health literacy
* Individuals with positive attitude towards dental health and dentist are attentive towards their oral health.

DETAILED DESCRIPTION:
This study will be conducted in two stages. The first stage includes a baseline cross-sectional investigation. Oral health literacy level will be assessed by conducting a structured interview. Background variables, attitude, socioeconomic factors and psychological factors shall be assessed using self-administered questionnaires. A clinical examination will be conducted including general health information and extended oral health examination. The oral health examination performed includes record of oral hygiene status such as dental caries and periodontal status. An assessment of oral bacteria will also be performed.

The second stage will be carried out approximately 6 months after starting with the baseline investigation. At that time a modified version of the questionnaires will be used followed by a shorter clinical examination. The modified questionnaires at the second data collection exclude some background variables. The clinical examination carried out during this time will be on dental plaque and bleeding index and the level of oral bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Participants > 20 years of age.
* Participants who master the Norwegian language.
* Participants who are registered at the university dental clinic (IKO).

Exclusion Criteria:

* People who do not master the Norwegian language.
* Strongly visually impaired people that have difficulty in reading.
* People with a history of heart-attack in the past 6 months.
* Immune- compromised people and organ- transplanted people.
* People with other conditions that might lead to more disadvantages than advantages by participating

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan O Bergdahl, Professor, Principal Investigator — University of Tromsoe, Norway
Locations (2):
- Norway (2):
  - Institute of Clinical Dentistry, University of Tromsø, Tromsø
  - Public Dental Service Competence Centre of Northern Norway (TkNN), Tromsø

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the waiting list at Tromsø University Dental Clinic. The recruitment started in May 2010 after approval from the regional ethical committee. Information letter with consent form was provided.
Pre-assignment Details: Enrolled participants:
  Total excluded n=46
  * Not meeting the inclusion criteria (n=11)
  * Declined to participate (n=35)
Groups:
- Experiment: Communication Adapted to Health Literacy Level: Participants in the experimental group got individualized communication regarding their oral health. The communication was adapted to the measured Health Literacy level of each participant. Health Literacy communication theory was utilized in order to adapt the communication to the participants Health literacy level. Two-way communication with use of models, illustrative pictures and teach-back method was emphasized. Up to 30 minutes was available for this intervention conversation.
- Control: Short Standard Information: Participants in the control group got short standard information after the clinical measurement, as usual in general dental clinical practice. E.g. If there was gingival bleeding, participants got a message that their gums were bleeding and that dental floss was recommended.
Period: Overall Study
Arm/Group | Experiment: Communication Adapted to Health Literacy Level | Control: Short Standard Information
Started | 64 | 69
Completed | 62 | 64
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Individualized Oral Health Instruction: Individualized oral health instruction adapted to the patients oral health literacy level
- Ordinary Oral Health Instruction: Oral health instruction commonly used in general practice
- Total: Total of all reporting groups
Arm/Group | Individualized Oral Health Instruction | Ordinary Oral Health Instruction | Total
Number analyzed (Participants) | 64 | 69 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 63 | 117
  >=65 years | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (15.19) | 46.4 (14.23) | 47.9 (14.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 76
  Male | 25 | 32 | 57
Region of Enrollment [Number; unit: participants]
  Norway | 64 | 69 | 133
health literacy level [Number; unit: paticipants]
  Inadequate health literacy | 15 | 24 | 39
  Marginal health literacy | 36 | 25 | 61
  Adequate health literacy | 13 | 20 | 33

OUTCOME MEASURES:

1. Primary Outcome: Gingival Index
Description: The gingival index of the individual was obtained by adding the values of each tooth (an average of 4 scores) and dividing by number of teeth examined with the resulting scores as follows 0.1-1.0 = mild inflammation; 1.1-2.0 = moderate inflammation; 2.1-3.0 = severe inflammation. The GI reference is Löe and Silness, 1963.
Time Frame: 6 months after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individualized Oral Health Instruction | Ordinary Oral Health Instruction
Number analyzed (Participants) | 64 | 69
units on a scale | 0.7190 (0.41599) | 1.1152 (0.45838)

2. Secondary Outcome: Plaque Index
Description: The plaque index of the individual was obtained by adding the values of each tooth (an average of 4 scores) and dividing by number of teeth examined with the resulting scores as follows 0.1-1.0 = low accumulation of plaque; 1.1-2.0 = Moderate accumulation of plaque; 2.1-3.0 = high accumulation of plaque.
  The Plaque index reference is Silness and Löe, 1964.
Time Frame: 6 months after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Individualized Oral Health Instruction; Ordinary Oral Health Instruction: The effect of intervention is evaluated using measures of plaque index
Arm/Group | Individualized Oral Health Instruction | Ordinary Oral Health Instruction
Number analyzed (Participants) | 64 | 69
units on a scale | 0.0805 (0.12958) | 0.3386 (0.34694)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Individualized Oral Health Instruction: The oral health instruction is individualized according to the patients oral health literacy level
- Control: The oral health instruction is according to standard clinical practice
Arm/Group | Individualized Oral Health Instruction | Control
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/69
Other Adverse Events (participants affected / at risk) | 0/64 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No